CLINICAL TRIAL: NCT05929885
Title: A Phase II Study of Metronomic Capecitabine, Oxaliplatin and UGT1A1 Genotype-directed Irinotecan in Metastatic Pancreatic Cancer Patients.
Brief Title: Metronomic Capecitabine, Oxaliplatin and UGT1A1 Genotype-directed Irinotecan in Metastatic Pancreatic Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LDOXIRI-PDAC-01
Record Dates: First submitted 2023-04-24; First posted 2023-07-03 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Low Dose OXIRI (LDOXIRI); Pancreatic Cancer; Irinotecan; Oxaliplatin; Capecitabine; Pharmacokinetics; Metronomic Chemotherapy; UGT1A1
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 43 patients will be enrolled in two stages - In stage 1, a total of 19 patients will be recruited and evaluated for response and toxicity. In stage 2, another 24 patients will be recruited for further evaluation of response and toxicity. Up to 7 patients will be recruited to account for any drop outs (i.e. up to total of 50 patients).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Dose OXIRI (LD-OXIRI) (Experimental): Low Dose OXIRI (LD-OXIRI) regimen comprises Metronomic Oxaliplatin (O) and Metronomic Capecitabine (xeloda; X) in combination with UGT1A1-directed dosing of Irinotecan (IRI).
  Interventions: Drug: Low Dose OXIRI (LD-OXIRI)

INTERVENTIONS:
Drug: Low Dose OXIRI (LD-OXIRI) — The LD-OXIRI regimen will be administered in the following sequence:
  * metronomic capecitabine (Xeloda; X) 650mg/m2 will administered twice a day on a daily a continuous basis;
  * intravenous metronomic oxaliplatin (O) 50 mg/m2 will be infused over 120 minutes on days 1 and 8 of a 21 day-cycle; followed by
  * intravenous irinotecan (I) will be infused over 90 minutes on days 1 and 8 of a 21 day-cycle. The dose of irinotecan will be based on the particular patient's UGT1A1*6 and UGT1A1*28 genotype status.

SUMMARY:
This is a single-centre, non-randomized, open label phase II trial to be conducted at the National Cancer Centre, Singapore (NCCS). Patients diagnosed with metastatic PDAC will be eligible to enrol.

The investigators hypothesize the anticancer activity of low dose OXIRI (LD-OXIRI) regimen comprising of metronomic oxaliplatin (O) and metronomic capecitabine (xeloda; X) in combination with UGT1A1-directed dosing of irinotecan (IRI) to be a tolerable regimen in patients with advanced PDAC and will lead to a favourable response rate.

Patients will be prospectively enrolled in two stages - In stage 1, patients will be recruited and evaluated for response and toxicity. In stage 2, more patients will be recruited for further evaluation of response and toxicity.

DETAILED DESCRIPTION:
Eligible patients will be recruited from the National Cancer Centre, Singapore (NCCS). Patients will be referred for assessment by the primary physician to a study investigator for screening. Informed written consent for entry into the trial will be obtained from the patient by a delegated investigator.

All patients eligible for study entry will receive the LD-OXIRI regimen at the National Cancer Centre, Singapore. All concomitant medication taken during the study must be recorded. If a drug is administered prophylactically, this must be noted. The patients will not receive any other investigational drugs while on this study.

There will be a screening period of 28 days, a treatment period till disease progression or unacceptable toxicity, and a post-treatment follow up period of up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

The patient must meet all of the inclusion criteria to participate in the study.

1. Aged above 21
2. Histopathological diagnosis of pancreatic cancer
3. Advanced disease not amenable to curative resection (locally advanced or metastatic disease)
4. Measureable disease by RECIST 1.1 criteria
5. Life expectancy of at least 12 weeks
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
7. Adequate hematologic function (granulocyte count ≥ 1.5 × 10**9/L, platelet count ≥ 100 × 10**9/L),
8. Adequate hepatic function (total bilirubin ≤ 1.5 x the upper limits of normal [ULN], AST and ALT, ALP ≤ 3 x ULN or < 5 x ULN in case of hepatic involvement),
9. Adequate renal function (creatinine clearance > 50 mL/min) will be eligible for inclusion into the study.
10. Able to provide written and informed consent

Exclusion Criteria:

Any patient meeting any of the exclusion criteria at baseline will be excluded from participation.

1. History of another malignancy within 5 years prior to registration. Patients with a past history of adequately treated carcinoma-in-situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and superficial transitional cell carcinoma of the bladder are eligible. Patients with a history of other malignancies are eligible if they have been continuously disease free after definitive primary treatment for at least 5 years.
2. Untreated CNS metastases or leptomeningeal disease. Patients with brain metastases that have been treated, and are asymptomatic, and have been stable for 3 or more months after treatment are allowed. A baseline CT or MRI brain is only required if there is clinical suspicion of CNS involvement.
3. Concurrent illness, including severe infection, that may jeopardise the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety
4. Serious medical or psychiatric conditions that might limit the ability of the patient to comply with the protocol
5. Treatment with palliative chemotherapy or radiotherapy within 4 weeks prior to enrolment into the study
6. Major surgery within two weeks prior to enrolment into the study
7. Patients on chronic immunosuppressive therapy
8. Pregnancy, lactation or inadequate contraception. Women of childbearing potential must have a negative pregnancy test within 3 days of enrolment and agree to use a reliable means of contraception. Men must have been surgically sterilised or agree to use a barrier method of contraception
9. Patients on anticoagulant therapy with vitamin K antagonists.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR). | Up to 3 years.
  The proportion of patients who have a partial or complete response as specified in RECIST 1.1.
Clinical Benefit Rate (CBR). | Up to 3 years.
  The percentage of advanced cancer patients who achieve complete response, partial response, or at least six months of stable disease as specified in RECIST 1.1.
The Grade 3-5 Toxicity Rate. | Up to 3 years.
  The proportion of patients who have adverse event(s) with Grade 3-5 toxicity as defined in CTCAE 5.0.

SECONDARY OUTCOMES:
Maximum plasma concentration [(Cmax)] of low dose Capecitabine and its intermediary metabolites (5'-deoxy-5-fluorocytidine [DFCR] and 5'- deoxy-5-fluorouridine [DFUR]) and 5FU. | At predose, 1 hr, end of irinotecan infusion on Cycle 1 Day 1 (each cycle is 21 days)
  Maximum plasma concentration [(Cmax)] of low dose capecitabine and its intermediary metabolites (5'-deoxy-5-fluorocytidine [DFCR] and 5'- deoxy-5-fluorouridine [DFUR]) and 5FU at Cycle 1 Day 1.
Trough concentration of low dose capecitabine and its intermediary metabolites and 5FU. | At predose of Cycle 2 Day 1 and Cycle 3 Day 1 (each cycle is 21 days)
  Trough concentration of low dose capecitabine and its intermediary metabolites (5'-deoxy-5-fluorocytidine [DFCR] and 5'- deoxy-5-fluorouridine [DFUR]) and 5FU.
Immunophenotyping from extracted peripheral blood mononuclear cells (PBMCs) - measurement of cytokine and chemokine concentrations in picograms per milliliters using multiplex flow cytometry. | Up to 3 years.
  Immunophenotyping from extracted peripheral blood mononuclear cells (PBMCs) - measurement of cytokine and chemokine concentrations in picograms per milliliters using multiplex flow cytometry at these time-points: at predose, end of oxaliplatin infusion, end of irinotecan infusion on Cycle 1 Day 1 (each cycle is 21 days); at predose of Cycle 2 Day 1 and at disease progression (up to three years).
Genomic analysis of circulating tumour DNA (ctDNA). | Up to 3 years.
  Genomic analysis of circulating tumour DNA (ctDNA) from whole blood at these time-points: at predose of every two cycles (Cycle 1 Day 1, Cycle 3 Day 1, Cycle 5 Day 1, etc - each cycle is 21 days) and at disease progression (up to three years).
Identification of exosomal proteins secreted by extracellular vesicles from plasma. | Up to 3 years.
  Identification of exosomal proteins secreted by extracellular vesicles from plasma using mass spectrometry, at the following time-points: at predose, end of oxaliplatin infusion, end of irinotecan infusion on Cycle 1 Day 1 (each cycle is 21 days); at predose of Cycle 2 Day 1 and at disease progression (up to three years).
Progression-free survival (PFS). | Up to 3 years.
  Time from first dose of treatment to disease progression or death, whichever comes first.
Overall survival (OS). | Up to 3 years.
  Time from first dose to death.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Joycelyn LEE, MBBS, MRCP (UK), M Med, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No